CLINICAL TRIAL: NCT03625947
Title: Prospective, Observational Study on the Efficacy, the Safety and the Predictors of Success of Argon Plasma Coagulation in the Treatment of Patients With Hemoptysis Caused by Endobronchial Malignancies
Brief Title: Efficacy and Safety of Argon Plasma Coagulation in the Treatment of Patients With Hemoptysis Caused by Endobronchial Malignancies
Status: Terminated | Type: Observational
Why Stopped: Recruitment issues during pandemic (2020-2021)
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Michele Mondoni, Principal investigator, University of Milan
Other Study IDs: Argon
Record Dates: First submitted 2018-07-29; First posted 2018-08-10 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hemoptysis; Cancer
Keywords: Hemoptysis; Lung cancer
MeSH Terms: conditions — Hemoptysis; Neoplasms; Lung Neoplasms | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemoptysis patients: Hemoptysis patients caused by endobronchial malignancies
  Interventions: Other: Argon Plasma Coagulation

INTERVENTIONS:
Other: Argon Plasma Coagulation — Patients will be treated with Argon Plasma Coagulation. Argon plasma coagulation (APC) is a form of non contact electrocoagulation. APC utilizes electrically conductive argon plasma as a medium to deliver high-frequency current via a flexible probe. The argon plasma flow transfers electricity between the probe and the target tissue. Tracheobronchial access is obtained by passing the probe through the working channel of the bronchoscope. On arrival to the tissue, the application of energy causes uniform zones of desiccation, coagulation and devitalization in the areas receiving treatment, thus inducing hemostasis.
  Other Names: APC

SUMMARY:
The aim of this study is to evaluate the efficacy, the safety and the main predictors of success of bronchoscopic Argon Plasma Coagulation in patients with hemoptysis caused by endobronchial malignancies.

DETAILED DESCRIPTION:
Hemoptysis is a challenging symptom which may be frequently related to endobronchial malignancies. Patients with central neoplasms and hemoptysis show a lower median survival than patients with no bleeding and endobronchial neoplasms and/or patients with hemoptysis and peripheral malignant lesions.

Hemoptysis control without recurrence at 48 hours after bronchoscopic interventions may improve survival in patients with mild bleeding and endobronchial malignancies.

Argon Plasma Coagulation is considered one of the most effective techniques for endobronchial management of hemoptysis in this subset of patients. Nevertheless, few data are available in literature on its efficacy and safety, and the main predictors of success are still unclear.

In this prospective, observational study, investigators aim to evaluate the efficacy (i.e. immediate bleeding cessation without recurrence during the following 48 hours) of endoscopic Argon Plasma Coagulation in patients with hemoptysis caused by endobronchial neoplasms.

Investigators will also evaluate the safety of the procedure, the main variables associated to a successful intervention, the presence of hemoptysis relapses and patients overall survival to 3,5 months after the bronchoscopic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hemoptysis caused by endobronchial (i.e. identifiable with flexible bronchoscopy) malignancies, without coagulopathy or other medically correctable causes of bleeding, who need endoscopic intervention with Argon Plasma Coagulation to stop bleeding
* Adult patients who are able to tolerate bronchoscopy
* Adult patients who are able to sign the written informed consent for the study participation

Exclusion Criteria:

* Patients with hemoptysis caused by endobronchial malignancies with coagulopathy or other medically correctable causes of bleeding.
* Patients who are not able to tolerate bronchoscopy
* Patients with hemoptysis without identifiable endobronchial malignancies during flexible bronchoscopy
* Patients with Pace-Maker and/or Automated Implantable Cardioverter- Defibrillator(AICD)
* Patients who refuse/are not able to sign the informed consent for the study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hemoptysis caused by endobronchial malignancies who need an endoscopic intervention (i.e Argon Plasma Coagulation) to stop the bleeding
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with bleeding cessation without recurrence at 48 after bronchoscopic Argon Plasma Coagulation | 48 hours
  Percentage of patients with bleeding cessation without recurrence at 48 hours after bronchoscopic Argon Plasma Coagulation employed to stop hemoptysis caused by endobronchial malignancies

SECONDARY OUTCOMES:
Incidence of adverse events | 48 hours
  Incidence of adverse events following bronchoscopic Argon Plasma Coagulation in the treatment of patients with hemoptysis and endobronchial malignancies
Incidence of hemoptysis recurrences | 3,5 months
  Incidence of hemoptysis recurrences (number of relapses)
Number of patients with hemoptysis and endobronchial malignancies who are still alive at the end of the follow-up | 3,5 months
  Number of patients with hemoptysis and endobronchial malignancies who are still alive after 3,5 months after the endoscopic intervention
Clinical and endoscopic factors (composite measure) associated to bleeding cessation after the intervention | 48 hours
  Clinical and endoscopic factors (composite measure) associated to bleeding cessation after the intervention (i.e. age, gender, ethnicity, smoking history, cancer type and stage, ECOG performance Status, concomitant heart, lung, kidney and liver disease, antiplatelet/anticoagulant therapy, creatinine and hemoglobin level and platelet count, PT and PTT values; endoscopic location of malignancy (i.e. lobe and side), endoscopic growth pattern of malignancy (i.e. exophytic, submucosal/peribronchial growth), current/former chemotherapy and radiation therapy on the chest, time from malignancy diagnosis to hemoptysis onset, time from hemoptysis onset to endoscopic treatment, necessity of blood transfusion).

CONTACTS AND LOCATIONS:
Overall Officials: Michele Mondoni, MD, Principal Investigator — University of Milan
Locations (1):
- Michele Mondoni, Milan, Italy